CLINICAL TRIAL: NCT01026285
Title: Observational, Non-interventional Registry to Assess Medication Usage Patterns in Clinical Routine Practice, in Subjects Receiving Antipsychotic Treatment With Risperidone Long Acting Injectable (Gluteal or Deltoid) or Oral Antipsychotics
Brief Title: InORS - International Observational Registry on Schizophrenia With Injectable Risperidone and Oral Antipsychotics
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016630; RISSCH4230 (Other: Janssen-Cilag International NV, Belgium)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Risperdal Consta
MeSH Terms: conditions — Schizophrenia | interventions — Antipsychotic Agents

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- antipsychotic treatment: Risperidone Long-Acting injectable or oral antipsychotics According to label
  Interventions: Drug: Risperidone Long-Acting injectable or oral antipsychotics

INTERVENTIONS:
Drug: Risperidone Long-Acting injectable or oral antipsychotics — According to label

SUMMARY:
International Observational Registry on Schizophrenia

DETAILED DESCRIPTION:
This is an observational, non-interventional registry designed to assess medication usage patterns and to explore, in clinical routine practice, long-term outcomes and relevant factors for patient adherence to treatment, in patients receiving antipsychotic treatment with risperidone long-acting injectable (RLAI) or oral antipsychotics. Six month retrospective data and 1 year prospective data will be collected. According to label

ELIGIBILITY:
Inclusion Criteria:

* Patients must satisfy the following criteria to be eligible for documentation in this non-interventional study: Diagnosis of schizophrenia as well as 6 months of retrospective clinical records
* Newly initiated on or switched to RLAI or an oral antipsychotic treatment (either atypical or conventional), not longer than 2 weeks ago
* Signed informed consent (either signed by the patient or his/her legal representative) is available at the beginning of documentation
* any schizophrenic patient (including those for whom a legal representative must sign consent) can be involved in the study

Exclusion Criteria:

* Established treatment refractory schizophrenia, defined as treatment failures with adequate trials (adequate as judged by the treating physician) of more than 2 second generation (atypical) antipsychotics and/or clozapine
* History of neuroleptic malignant syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 1085 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
prospectively assess medication usage patterns under routine clinical practice related to initiation of treatment with risperidone RLAI and oral antipsychotic treatments | baseline, month 1, 3, 6, 9 & 12

SECONDARY OUTCOMES:
To collect 6-month retrospective and 1-year prospective data to allow the exploration of treatment outcomes including hospitalizations and rehospitalizations, with RLAI and oral antipsychotics, in relation to previous treatments | 1, 3, 6, 9, 12 month
To evaluate the reasons for initiation and/or discontinuation of new antipsychotic medications, including patient satisfaction with treatment | 1, 3, 6, 9, 12 month
To explore relevant factors for patient adherence to treatment | 1, 3, 6, 9, 12 month
To document clinical effectiveness and functionality of patients on RLAI and oral antipsychotics in daily clinical practice (as measured by the Global Assessment of Functioning [GAF] scale | 1, 3, 6, 9, 12 month
Long-term safety data of RLAI (25, 37.5 or 50 mg every 2 weeks) and oral antipsychotics will be collected | 1, 3, 6, 9, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (98):
- Czechia (6):
  - Brno
  - České Budějovice
  - Most
  - Olomouc
  - Prague
  - Přerov
- France (20):
  - Bar-le-Duc
  - Boulogne-Billancourt
  - Bourg-en-Bresse
  - Challans
  - Créteil
  - Dax
  - La Roche-sur-Yon
  - La Seyne-sur-Mer
  - Laxou
  - Marseille
  - Mont-Saint-Martin
  - Montpellier
  - Morlaix
  - Plouguernével
  - Rennes
  - Saint-Avé
  - Saint-Égrève
  - Sarreguemines
  - Verdun
  - Villejuif
- Germany (40):
  - Augsburg
  - Bad Honnef
  - Berlin
  - Bochum
  - Butzbach
  - Chemnitz
  - Coesfeld
  - Cologne
  - Dortmund
  - Dresden
  - Düsseldorf
  - Ebensfeld
  - Frankfurt
  - Fürth
  - Geithain
  - Greifswald
  - Grevenbroich
  - Hamburg
  - Ilmenau
  - Köthen
  - Krefeld
  - Leipzig
  - Limburg
  - Löhne
  - Magdeburg
  - Mannheim
  - München
  - Neuss
  - Oranienburg
  - Plauen
  - Potsdam
  - Riesa
  - Schleswig
  - Stolberg
  - Stralsund
  - Ulm
  - Velbert
  - Wetzlar
  - Wismar
  - Wuppertal
- Greece (8):
  - Arta
  - Athens
  - Chania
  - Crete
  - Ioannina
  - Larissa
  - Thessalonikis
  - Véroia
- Russia (4):
  - Kronshtadt
  - Nizhny Novgorod
  - Saint Petersburg
  - Yekaterinburg
- South Africa (2):
  - Birmingham, AL
  - Pretoria
- Spain (8):
  - A Coruña
  - Burgos
  - Getafe
  - Madrid
  - Monforte de Lemos
  - Salamanca
  - Valladolid
  - Vigo
- Turkey (Türkiye) (10):
  - Adana
  - Ankara
  - Erzurum
  - Eskişehir
  - Istanbul
  - Izmir
  - Kocaeli
  - Manisa
  - Mersin
  - Trabzon

REFERENCES:
- See also: InORS - International Observational Registry on Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=227&filename=CR016630_CSR.pdf